CLINICAL TRIAL: NCT04658212
Title: A Multicenter Randomized Controlled Study of 3D Laparoscopy Versus Endoscopy in the Treatment of Choledocholithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSBS-LSES-1
Record Dates: First submitted 2020-11-21; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Choledocholithiasis; ERCP
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D LCBDE group (Experimental)
  Interventions: Procedure: 3D LCBDE
- ERCP group (Active Comparator)
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: 3D LCBDE — three-dimensional (3D) video system for LCBDE (laparoscopic cholecystectomy and laparoscopic common bile duct exploration )
  Arms: 3D LCBDE group
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography (ERCP)
  Arms: ERCP group

SUMMARY:
The incidence of choledocholithiasis is gradually rising with the increase of gallstone incidence. The popular minimally invasive treatment options include endoscopic retrograde cholangiopancreatography (ERCP) and laparoscopic common bile duct exploration (LCBDE). Currently, three-dimensional (3D) video system for laparoscopy is developed to ofer surgeon a superior depth perception and a much better user experience, thus potential increasing operation accuracy and stability. It have suggested that compared with 2D laparoscopy, 3D laparoscopy can effectively reduce operation time and numbers of errors. However, rare experimental studies are performed to evaluate the safety and effectiveness of 3D laparoscopy in choledocholithiasis patients. The aim of this study is to compare the perioperative outcomes between 3D laparoscopy and ERCP in choledocholithiasis patients through a multicenter randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of choledocholithiasis based on preoperative image studies including abdominal ultrasonography, computed tomography (CT), and/or magnetic resonance cholangiopancreatography (MRCP) with relevant supporting laboratory examinations
2. Age <80y and >18y
3. Non-emergency surgery

Exclusion Criteria:

1. Diagnosis of Mirizzi's syndrome,
2. Acute suppurative cholangitis
3. Detection of bilioenteric anastomosis
4. Pathological diagnosis of cholangiocarcinoma
5. Extended surgery due to multiple biliary strictures,
6. Intrahepatic stones

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative Complication Rate | 1 month after surgery

IPD SHARING:
Plan to Share IPD: No